CLINICAL TRIAL: NCT00280488
Title: Enhanced MI With Alcohol Positive Trauma Patients
Brief Title: Enhanced Motivational Interviewing With Alcohol Positive Trauma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Peter Monti, Ph.D., Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAMON-009892-11A1; 3R01AA009892-15S1 (NIH); NIH grant AA009892-11A1
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Alcohol Abuse; Alcohol Dependence
Keywords: Motivational Interviewing; Alcohol Abuse; Alcohol Dependence; Emergency Care Setting
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1) MI with SO (Active Comparator): Motivational Interviewing (MI), a brief, directive, non-confrontational intervention, with inclusion of a significant other (SO) in prolonged, intensive alcohol treatment.
  Interventions: Behavioral: Motivational Interview
- 2) MI with patient only (Active Comparator): Motivational Interviewing (MI), a brief, directive, non-confrontational intervention, with the individual patient
  Interventions: Behavioral: Motivational Interview
- 3) Assessment only (Active Comparator): In the assessment-only condition, patients will receive only assessment of their drinking at baseline.
  Interventions: Behavioral: Assessment

INTERVENTIONS:
Behavioral: Motivational Interview — Two intervention sessions timed to occur in the hospital, and 1 booster session, occurring 1 month following discharge.
  Arms: 2) MI with patient only
Behavioral: Assessment — In the assessment-only condition, patients will receive only assessment of their drinking at baseline.
  Arms: 3) Assessment only
Behavioral: Motivational Interview — Two intervention sessions timed to occur in the hospital, and 1 booster session, occurring 1 month following discharge.
  Arms: 1) MI with SO

SUMMARY:
The primary goal of this study is to test the efficacy of a brief intervention that includes the patient and a significant other, relative to an intervention including the patient only, for reducing alcohol use and alcohol-related problems among trauma patients.

DETAILED DESCRIPTION:
Alcohol-positive trauma patients are more likely to be readmitted to a trauma center or subsequently die from an injury than are alcohol-negative patients. Empirically supported treatments to reduce alcohol use and alcohol-related problems (e.g., injuries, drinking and driving) in this high-risk population are needed, but few exist. This randomized controlled clinical trial assesses the efficacy of a brief intervention that includes the patient and a significant other, relative to an intervention including the patient only, for reducing alcohol use and alcohol-related problems among trauma patients.

Motivational Interviewing (MI), a brief, directive, non-confrontational intervention, has demonstrated some promise in this setting. Further, inclusion of a significant other (SO) in prolonged, intensive alcohol treatment appears to improve treatment retention and efficacy. Although inclusion of an SO in MI has been suggested, there are few data to support this endorsement.

Accordingly, this study will address whether motivational interviewing including both the trauma patient and an SO can more effectively decrease and maintain reductions in alcohol use and alcohol-related problems 6 and 12 months following discharge from the trauma unit than MI with the individual patient or an assessment-only condition.

The 2 MI groups will each receive 2 intervention sessions timed to occur in the hospital, and 1 booster session, occurring 1 month following discharge.

In the assessment-only condition, patients will receive only assessment of their drinking at baseline. This proposal will allow us to address the next phase of our program of research designed to develop easily disseminable treatments for these high-risk populations in medical settings. This study will also address potential mediators (motivation to change alcohol use, self-efficacy, alcohol treatment attendance, and social support for abstinence) and moderators of MI effects. The cost-effectiveness of the intervention will also be addressed.

Thus, this study will address both a significant public health problem and provide important information about MI mechanisms that may be relevant to the broader addiction treatment community.

ELIGIBILITY:
Inclusion Criteria:

* admitted to trauma unit
* greater than 18 years old
* had a blood alcohol concentration (BAC) greater than .01% according to a biochemical test OR self-reported drinking alcohol in the 6 hours prior to the event that caused their hospital visit OR scored 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT)
* identify at least one eligible significant other

Exclusion Criteria:

* not English-speaking
* had a self-inflicted injury
* in police custody
* did not pass a mental status exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-05; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 12 months
Alcohol-related problems (e.g., drinking and driving) | 12 months

SECONDARY OUTCOMES:
Cost-effectiveness of intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Monti, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - Brown University, Providence, Rhode Island